CLINICAL TRIAL: NCT04332042
Title: TOFAcitinib in Patients With Early Onset SARS-CoV2 Interstitial Pneumonia
Brief Title: TOFAcitinib in SARS-CoV2 Pneumonia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Armando Gabrielli, Full Professor Internal Medicine, Università Politecnica delle Marche
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOFACoV
Record Dates: First submitted 2020-03-28; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: SARS-COv2 Related Interstitial Pneumonia
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Intervention Model Description: prospective cohort study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tofacitinib (Experimental): Tofacitinib cp 5mg: 2pills twice a day for 14 days
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Tofacitinib 10mg twice a day will be administered within 24h from hospital admission for 14 days

SUMMARY:
Immune-mediated lung injury plays a pivotal role in severe interstitial pnemumonia related to SARS-CoV2 infection. Tofacitinib, a JAK1/3-Inhibitor, could mitigate alveolar inflammation by blocking IL-6 signal. The aim of this prospective single cohort open study is to test the hypotesis that early administration of tofacitinib in patients with symptomatic pneumonia could reduce pulmonary flogosis, preventing function deterioration and the need of mechanical ventilation and/or admission in intensive care units.

DETAILED DESCRIPTION:
Interstitial Pneumonia is the main complication of SARS-CoV2 infection. Immune system hyperactivation, leading to alveolar inflammation, is the main mechanism in determining lung damage. Evidence are accumulating about the pivotal role played by IL-6 in this disease. Preliminary evidence, indeed, point out the efficacy of an IL-6 receptor inhibitor in improving clinical conditions in a proportion of rapidly deteriorating patients. Our hypotesis is that a precocious inhibition of IL-6 signal, by the administration of tofacitinib (JAK 1/3 Inhibitor), could hinder the progression to more severe grades of lung inflammation leading to pulmonary function deterioration. In a prospective single cohort open study, 50 patients admitted in Hospital due to SARS-CoV 2 symptomatic interstitial pneumonia, but not requiring mechanical ventilation, will be enrolled. Tofacitinb will be administered every day for 14 days, starting within 24 h from the admission. The primary outcome is to evaluate the effect of this drug on the rate of patients who will need mechanical ventilation. Safety in this population will also be actively monitored.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV2 Infection diagnosed by rt-PCR
* Rx or CT-scan confirmed interstitial pneumonia
* Hospital admission from less than 24h
* Written Informed Consent

Exclusion Criteria:

* Age <18 ys or >65
* Patients in mechanical ventilation at time of admission
* Severe Hearth failure (NYHA 3 or 4)
* Severe History of Chronic Ischemic Hearth Disease, defined as history of Major Adverse Cardiovascular Event and/or recent (one year) revascularization.
* History of recurrent Deep Venous Thrombosis and Pulmonary Embolism
* Active Bacterial or Fungal Infection
* Hematological cancer
* Metastatic or intractable cancer
* Pre-existent neurodegenerative disease
* Severe Hepatic Impairment
* Severe Renal Failure (Creatinine Clearance <30ml/h)
* Active Herpes zoster infection
* Severe anemia (Hb<9g/dl)
* Lymphocyte count below 750/mcl
* Neutrophil count below 1000/mcl
* Platelet count below 50000/mcl
* Pregnancy or Lactation
* Inability to give informed consent (severe transitory or permanent mental impairment, incapacitation)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04-10 (Estimated); Primary Completion 2020-06-20 (Estimated); Study Completion 2020-07-10 (Estimated)

PRIMARY OUTCOMES:
need of mechanical ventilation | day 14
  Rate of patients needing mechanical ventilation to maintain PaO2/FIO2>150 or, if PaO2 data not available, to maintain SO2>94% with FiO2 0,5.

SECONDARY OUTCOMES:
need of admission in intensive care unit | day 14
  Rate of patients needing admission to the intensive care unit for oro-tracheal intubation and/or evidence of Multiple Organ Disfunction
death | day 28
  rate of patients dead
rate of adverse events | day 28
  rate and type of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedali Riuniti di Ancona, Ancona, The Marches, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tian S, Hu W, Niu L, Liu H, Xu H, Xiao SY. Pulmonary Pathology of Early-Phase 2019 Novel Coronavirus (COVID-19) Pneumonia in Two Patients With Lung Cancer. J Thorac Oncol. 2020 May;15(5):700-704. doi: 10.1016/j.jtho.2020.02.010. Epub 2020 Feb 28. PMID 32114094
- [Background] Ashour HM, Elkhatib WF, Rahman MM, Elshabrawy HA. Insights into the Recent 2019 Novel Coronavirus (SARS-CoV-2) in Light of Past Human Coronavirus Outbreaks. Pathogens. 2020 Mar 4;9(3):186. doi: 10.3390/pathogens9030186. PMID 32143502
- [Background] Zumla A, Hui DS, Azhar EI, Memish ZA, Maeurer M. Reducing mortality from 2019-nCoV: host-directed therapies should be an option. Lancet. 2020 Feb 22;395(10224):e35-e36. doi: 10.1016/S0140-6736(20)30305-6. Epub 2020 Feb 5. No abstract available. PMID 32035018
- [Background] Rose-John S, Scheller J, Schaper F. "Family reunion"--A structured view on the composition of the receptor complexes of interleukin-6-type and interleukin-12-type cytokines. Cytokine Growth Factor Rev. 2015 Oct;26(5):471-4. doi: 10.1016/j.cytogfr.2015.07.011. Epub 2015 Jul 6. No abstract available. PMID 26235233
- [Background] McInnes IB, Byers NL, Higgs RE, Lee J, Macias WL, Na S, Ortmann RA, Rocha G, Rooney TP, Wehrman T, Zhang X, Zuckerman SH, Taylor PC. Comparison of baricitinib, upadacitinib, and tofacitinib mediated regulation of cytokine signaling in human leukocyte subpopulations. Arthritis Res Ther. 2019 Aug 2;21(1):183. doi: 10.1186/s13075-019-1964-1. PMID 31375130